CLINICAL TRIAL: NCT02822885
Title: Uterine Artery and Spiral Artery Doppler Parameters in Patients With Postmenopausal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, MD, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sleem
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Postmenopausal Bleeding
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasonography (Experimental): Ultrasonographic assessment of the thickness of the endometrium of the uterus and transvaginal color Doppler ultrasonography for measurements of Pulsatility index and resistance indices of uterine arteries and spiral arteries
  Interventions: Radiation: Ultrasonography

INTERVENTIONS:
Radiation: Ultrasonography — Ultrasonographic assessment of the thickness of the endometrium of the uterus and transvaginal color Doppler ultrasonography for measurements of Pulsatility index and resistance indices of uterine arteries and spiral arteries
  Other Names: color Doppler ultrasonography

SUMMARY:
This study was to investigate the diagnostic value of ultrasonography and blood flow measurements in uterine arteries and spiral arteries by transvaginal color Doppler ultrasonography in the detection of the endometrial pathology in women with postmenopausal bleeding.

DETAILED DESCRIPTION:
This prospective Cross-sectional Observational study will be conducted at the Department of Obstetrics and Gynecology, Banha University, Egypt during the period starting from January 2014. The study protocol will be approved by the Local Ethics Committee and written informed consent will be obtained from each patient before the study commenced.

Seventy patients with postmenopausal bleeding will be included in the study after verbal consent. They will be recruited from patients attending gynecologic clinic in Banha University hospital.

All patients will be subjected to the following:

For all included women the following will be done:

1. Full history taking.
2. Complete general, abdominal, and local examination.
3. Ultrasonographic assessment of the uterus

All data were performed for all patients in the lithotomy position after they had emptied their bladder using a 7.5 megahertz transducer by a single operator.

1. Using colour Doppler in the 2D mode, flow velocity waveforms were obtained from the ascending main branch of the uterine artery on the right and left side of the cervix in a longitudinal plane before they entered the uterus.
2. The gate of the Doppler was positioned when the vessel with good colour signals was identified on the screen. Pulsatility index of the uterine arteries were calculated electronically when similar consecutive waveforms of good quality were obtained and the averaged uterine PI.

   Pulsatility index (PI):

   This index, also known as the mean pulsatility index, to distinguish it from the peak to peak pulsatility index, is expressed by: PI= (S-D) / Mean Where S is the peak systolic velocity, D is the end diastolic velocity and velocity is the time averaged maximum velocity over the cardiac cycle (1).
3. Blood flow velocity waveforms were evaluated in the spiral arteries at the sub endometrial region that is within 1 mm of the originally defined myometrial-endometrial contour (2).

Histopathological diagnosis of endometrium obtained by biopsy is the gold standard for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Endometrial thickness ≥ 5 mm measured by two-dimensional transvaginal ultrasound.
2. Pap smear is negative for malignancy.

Exclusion Criteria:

1. Postmenopausal woman on hormon replacement therapy.
2. Trans-vaginal examination not possible (Vaginal stenosis or patient refusing trans-vaginal ultrasound).
3. Adnexal pathology.
4. General causes of bleeding e.g: Hemophilia , anticoagulation therapy

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Moharam A ABDEL HAEY, MD, Principal Investigator — Benha University; AHMED WALEED A Mrad, MD, Study Director — Benha University
Locations (1):
- Benha university hospitalا, Banhā, Alqalubia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dickey RP. Doppler ultrasound investigation of uterine and ovarian blood flow in infertility and early pregnancy. Hum Reprod Update. 1997 Sep-Oct;3(5):467-503. doi: 10.1093/humupd/3.5.467. PMID 9528912
- [Background] Ng EH, Chan CC, Tang OS, Yeung WS, Ho PC. Endometrial and subendometrial blood flow measured during early luteal phase by three-dimensional power Doppler ultrasound in excessive ovarian responders. Hum Reprod. 2004 Apr;19(4):924-31. doi: 10.1093/humrep/deh205. Epub 2004 Mar 11. PMID 15016770
- See also: Banha university — http://www.bu.edu.eg

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasonography
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
Age, Customized [Mean (Standard Deviation); unit: years] | 59.85 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Pulsatility Indices (PI) of Spiral Artery According to Histological Diagnosis
Description: Pulsatility index is a measure of the variability of blood velocity in a vessel, and was calculated as the difference between the peak systolic and end diastolic velocities divided by the mean velocity during the cardiac cycle. Higher values are indicative of increased vascular resistance
Time Frame: two weeks
Population: All patients(N=70) were subdivided according to histological diagnosis to A-Benign lesion (N=60)
  1. Endometrial polyp(N=17)
  2. Hyperplasia(N=28)
  3. Non-specific(N=15) B-Malignant lesion(N=10)
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
index
  endometrial polyp(n=17) | 1.08 (.33)
  endometrial Hyperplasia(n=28) | 1.22 (0.33)
  endometrialNon-specif lesions | 1.07 (0.3)
  all endometrial benign lesions | 1.14 (0.32)
  endometrial cancer(n=10) | 0.57 (0.09)
Statistical Analysis 1: Comparison: Ultrasonography; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

2. Primary Outcome: Resistive Indices (PI) of Spiral Artery According to Histological Diagnosis
Description: The primary outcome measure is spiral artery resistive index (RI) .In ultrasonography,it can be calculated from the peak systolic velocity and end diastolic velocity of blood flow and is calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity.lower values are better than higher values.
Time Frame: two weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
index
  endometrial polyp(n=17) | 0.62 (0.05)
  endometrial hyperplasia(n=28) | 0.68 (0.14)
  Non-specif endometrial lesions | 0.58 (0.07)
  all benig endometrial lesions | 0.64 (0.12)
  endometrial cancer(n=10) | 0.46 (0.03)
Statistical Analysis 1: Comparison: Ultrasonography; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

3. Primary Outcome: Uterine Artery Resistive Index According to Histological Diagnosis
Description: The primary outcome measures is uterine artery resistive index (RI) .In ultrasonography,it can be calculated from the peak systolic velocity and end diastolic velocity of blood flow and is calculated with the following formula: (peak systolic velocity - end diastolic velocity)/peak systolic velocity.lower values are better than higher values.
Time Frame: two weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
index
  endometrial polyp.(n=17) | 0.68 (0.12)
  endometrial hyperplasia.(n=28) | 0.79 (0.1)
  non specifi endometrial lesions. | 0.73 (0.15)
  all benign endometrial lesions. | 0.74 (0.13)
  endometrial cancer(n=10) | 0.51 (0.04)
Statistical Analysis 1: Comparison: Ultrasonography; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

4. Primary Outcome: Uterine Artery Pulsatility Index According to Histological Diagnosis
Description: as for outcome 1
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
index
  endometrial polyp | 0.94 (0.18)
  endometrial hyperplasia | 1.21 (0.31)
  un specific endometrial lesions | 0.88 (0.2)
  all benign endometrial lesions | 1.05 (0.29)
  endometrial cancer lesions | 0.65 (0.09)
Statistical Analysis 1: Comparison: Ultrasonography; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

5. Primary Outcome: Endometrial Thickness According to Histological Diagnosis
Description: Endometrial Thickness was assessed by measuring the trilaminar halo of the Endometrial Thickness by trans vaginal sonography
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Ultrasonography
Number analyzed (Participants) | 70
millimeter
  endometrial polyp | 18 (3.40)
  endometrial hyperplasia | 7.98 (1.8)
  un specific lesions | 9.56 (2.5)
  all benign lesions | 11.215 (5)
  endometrial cancer | 16.8 (3.4)
Statistical Analysis 1: Comparison: Ultrasonography; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — All included p-values are calculated from collected data and not threshold values for statical significance

ADVERSE EVENTS:
Arm/Group | Ultrasonography
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes